CLINICAL TRIAL: NCT00433277
Title: Autoimmunity in Retinitis Pigmentosa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Semmelweis University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: KMolnar
Record Dates: First submitted 2007-02-06; First posted 2007-02-09 (Estimated); Last update posted 2007-02-09 (Estimated); Status verified 2007-02

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

INTERVENTIONS:
Drug: twice-daily dosage with 0.5% cyclosporine-A eyedrops

SUMMARY:
Using local immune suppression, the trial seeks evidence for the hypothesis that autoimmunity plays a role in the pathomechanism of retinitis pigmentosa.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of retinitis pigmentosa

Exclusion Criteria:

* Cataract
* Extremely low ERG wave amplitude (less than 8% of normal)

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Zoltán Z. Nagy, M.D., Study Director — Semmelweis University, Dept. of Ophthalmology
Locations (1):
- Semmelweis University, Dept. of Ophthalmology, Budapest, Hungary